CLINICAL TRIAL: NCT00806091
Title: Functional Proteomics of Alveolar Macrophages
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Philip Diaz, Professor of Internal Medicine, Ohio State University
Other Study IDs: 2004H0102
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: COPD
Keywords: AM proteomes will be compared between smokers with and without COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood BAL fluid breathe condensation saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD subjects: healthy subjects

SUMMARY:
The purpose of this study is to obtain young white blood cells (monocytes) from the investigators donated blood for research into how these cells change into large, mature white blood cells (macrophages) and how smoking causes Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
Our research goal is to identify new targets and strategies to help care for patients with Chronic Obstructive Pulmonary Disease (COPD). COPD is a chronic airway inflammatory disorder characterized by a progressive loss of pulmonary function. Mononuclear phagocytes are known to be critically involved in both repair/remodeling and destructive events in COPD. Although smoking is the chief environmental risk factor for COPD, the molecular details responsible for the genesis and progression of smoking-mediated COPD require further investigation. In searching for new knowledge and research strategies for this challenging topic, we have made substantial progress in mononuclear phagocyte proteomics and laid the groundwork for this translational research of COPD.

ELIGIBILITY:
Inclusion Criteria:

* COPD, smoker
* COPD, non smoker

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: smokers with and without COPD, general population
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2004-07; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
to define AM's pathogenic pathways underlying the development of COPD | end of study

SECONDARY OUTCOMES:
to determine protein polymorphism(s) that impact genetic susceptibility to COPD | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Wu, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States